CLINICAL TRIAL: NCT00010504
Title: Pilot Study of Acupuncture in Fibromyalgia
Brief Title: Acupuncture in Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01 AT000004-01M; R01AT000004-01 (NIH); NCT00006338 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Fibromyalgia; Pain
Keywords: acupuncture; fibromyalgia; pain; analgesia
MeSH Terms: conditions — Fibromyalgia; Pain; Agnosia | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
Fibromyalgia is the second most common rheumatic disorder, affecting approximately 8-10 million persons in the U.S., and is characterized by widespread musculoskeletal pain and soft tissue tenderness upon examination. This study focuses on the use of acupuncture as a mode of therapy for fibromyalgia. The issues under examination are: 1) the optimal duration of treatment, 2) the independent and synergistic effects of needle placement and needle stimulation, and 3) appropriate control strategies. The proposal utilizes a randomized, blinded, sham-controlled design to achieve these aims. Subjects are randomly assigned to one of four groups: 1)active site with stimulation, 2) active site, without stimulation, 3) sham site with stimulation, and 4) sham site, without stimulation. All subjects will receive acupuncture at escalating frequency, beginning at once per week and ending at 3 times per week. This "forced titration" design allows for the detection of inter-subject differences in responsiveness to acupuncture, as well as the factors which may predict responsiveness (or lack thereof). Secondary goals of the study are to collect data on the mechanism, safety, and cost-effectiveness of acupuncture in fibromyalgia, and to determine the optimal outcome measures, for a full scale research clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Must be a resident of the Washington DC area.
* Having met ACR criteria for fibromyalgia.
* Continued widespread pain for more than 50% of days.
* Willing to limit the introduction of any new medications or treatment modalities for control of fibromyalgia symptoms during the 13 weeks of active treatment.
* Able to travel to acupuncture site up to 3 times per week.
* Capable of giving informed consent.

Exclusion Criteria:

* Knowledge of acupuncture sufficient to prevent "blinding" of the subject.
* Presence of a known coagulation abnormality that would prevent safe use of acupuncture.
* Presence of a concurrent autoimmune or inflammatory disease that causes pain.
* Routine daily use of narcotic analgesics or history of substance abuse.
* Participation in other concurrent therapeutic trials.
* Pregnant or nursing mothers.
* Disability insurance payments.
* Ongoing litigation related to fibromyalgia.
* Contraindication for the use of acetaminophen or ibuprofen.
* Any impairment, activity, or situation that in the judgement of the Study Coordinator would prevent satisfactory completion of the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Cupps, M.D., Study Director — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States